CLINICAL TRIAL: NCT01860027
Title: Reliability of Clinical Eye Movement Tests as Screening Devices for Reading Disabilities
Brief Title: Eye Movements and Reading Disabilities
Acronym: EOMRD
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Shelly Meese, Project Manager, Scripps Health
Other Study IDs: EOMRD
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Reading Disability; Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Children with reading disabilities: Children diagnosed with reading disabilities (age 7 to 13).
- Children with eye movement disorders: Children diagnosed with eye movement disorders (age 7 to 13).
- Control Group: Children with normal reading ability and normal eye movements (age 7 to 13.

SUMMARY:
The mechanism of the eye movement anomalies seen in dyslexic patients is not well defined. Some optometrists use observational eye movement tests as screening devices for dyslexia and advocate eye movement therapy as a treatment option for dyslexia. The reliability of the clinical eye movement tests and the efficacy of the eye movement therapies have not been determined.

Saccades are the fast eye movements that move our eyes from one word to the next when we read. The eye movement recordings from patients diagnosed with reading disorders, extra ocular muscle imbalances and control patients (no learning disability or eye movement disorder) will be analyzed and compared. The sensitivity and specificity of detecting reading disorders will be determined for the Visagraph III and the Readalyzer. Although these clinical tests are frequently used to diagnose saccadic inaccuracies and diagnose dyslexia in school aged children, the validity of these clinical screening tests has not been determined.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 7 to 13 (Must be in at least 2nd grade, but not higher than 8th grade) 2. Complete ophthalmic examination performed by a pediatric ophthalmologist and orthoptist.

  3. All ocular structures must be within normal limits. 4. Best corrected visual acuity must be equal to or better than 20/30 in each eye.

  5. Group 1:
  1. Children with a reading disability must be given the diagnosis by a clinical educational specialist, educational psychologist or neuro-behavioral psychologist.
  2. Children with a reading disability may not have any ophthalmic anomaly determined by testing as described above. This includes but is not limited to amblyopia, strabismus, nystagmus, or any organic disease.

     6. Group 2

  a. Eye movement disorder confirmed by testing by a pediatric ophthalmologist and/or orthoptist b. All other ocular structures must be within normal limits (including visual acuity).

  7. Group 3:
  1. No evidence of reading disability, attention deficit disorder or ocular anomaly, including eye muscle or movement disorder as specified above.

     Exclusion Criteria:
* 1. Myopia more than - 6.00 diopters (spherical equivalent) in either eye. 2. Hyperopia more than + 6.00 diopters (spherical equivalent) in either eye. 3. History of vision therapy or orthoptic treatment 4. Any ocular anomaly with the exception of eye movement disorder for group 2.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with reading disorders, eye movement disorders or control (normal reading and eyemovements)between the ages of 7 and 13 are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09-01 (Actual); Study Completion 2014-09-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of clinical eye movement devices | June 2014
  The primary analysis will be determining the sensitivity and specificity of the eye movement recording devices to recognize reading disorders. The sensitivity (true positive rate) of the eye movement recorders will be determined by the ability of each device to recognize children with reading disorders in Group 1. The specificity of the recorders will be determined by calculating the false positives in group 2 (eye movement disorders), and group 3 (control subjects).

SECONDARY OUTCOMES:
Comparison of eye movement characteristics amongst patients with reading disorders, eye movement abnormalities and control subjects. | June 2014
  The secondary analysis will be a study group comparison of eye movement results for each reading variable using an analysis of covariance (ANCOVA) model. The 6 calculated reading variables are listed below and will be individually compared amongst the three groups.
  i. Fixations / 100 words ii. Regressions / 100 words iii. Average span of recognition iv. Average duration of fixation v. Reading rate with comprehension vi. Grade level Efficiency

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Ostrow, MD, Principal Investigator — Scripps Clinic; Laura Kirkeby, Orthoptics, Study Director — Scripps Clinic
Locations (1):
- Scripps Clinic, San Diego, California, United States